CLINICAL TRIAL: NCT05337098
Title: Non-Nutritive Sweetener Consumption (Aspartame and Sucralose) and Glucose Homeostasis in Older Adults With Prediabetes
Brief Title: Non-Nutritive Sweetener Consumption and Glucose Homeostasis in Older Adults With Prediabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R21AG075344-01 (NIH)
Record Dates: First submitted 2022-03-04; First posted 2022-04-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Continuous Glucose Monitoring; Oral Glucose Tolerance; Insulin Sensitivity; Inflammatory Markers
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aspartame (Active Comparator): Controlled feeding study. Dosage of aspartame will follow 25% of the acceptable daily intake (equivalent to 12.5 mg/kg for aspartame). This amount represents 750 mg/day of aspartame for a 60 kg adult.
  Interventions: Other: Non-Nutritive Sweetener Intake and impact on glucose homeostasis
- Sucralose (Active Comparator): Controlled feeding study. Dosage of sucralose will follow 25% of the acceptable daily intake (equivalent to 1.25 mg/kg for sucralose). This amount represents 75 mg/day of sucralose for a 60 kg adult.
  Interventions: Other: Non-Nutritive Sweetener Intake and impact on glucose homeostasis
- No NNS (Sham Comparator): Controlled feeding study with no non-nutritive sweeteners.
  Interventions: Other: Non-Nutritive Sweetener Intake and impact on glucose homeostasis

INTERVENTIONS:
Other: Non-Nutritive Sweetener Intake and impact on glucose homeostasis — Provision of either aspartame, sucralose, or control with no non-nutritive sweeteners to a controlled feeding study to determine impacts on glucose homeostasis.

SUMMARY:
Animal and observational research in humans suggest that specific types of non-nutritive sweeteners (NNS) may impair glycemic control. However, whether NNS consumption impacts glucose homeostasis in middle-aged/older adults with prediabetes is unknown, and potential mechanisms by which this could occur have yet to be identified. The overall objective of this R21 proposal is to establish proof-of-concept for alterations in glucose homeostasis following intake of sucralose, but not aspartame, in middle-aged/older adults with prediabetes compared to a eucaloric diet with no NNS.

DETAILED DESCRIPTION:
Observational research has linked intake of non-nutritive sweeteners (NNS), which are consumed daily by ~50% of middle-aged/older U.S. adults, with increased risk of type 2 diabetes (T2D). This risk may be exacerbated by advancing age, which is associated with low-grade chronic inflammation and increased risk of T2D. Current T2D prevention recommendations related to NNS usage are unclear and confusing; use as an alternative to added sugar intake is suggested but long-term NNS use is discouraged despite minimal research to support this recommendation. Animal and observational human studies suggest detrimental effects of some NNS on glucose homeostasis. Longer-term human studies largely demonstrate null findings. Differences in study design and a lack of rigor in existing research contribute to inconclusive findings. In addition, NNS are often studied as a single entity yet types of NNS vary in their absorption and metabolism (e.g., the two most commonly consumed NNS, sucralose and aspartame). Whether NNS consumption impacts glucose homeostasis in middle-aged/older adults with prediabetes is unknown, and potential mechanisms by which this could occur have yet to be identified. The overall objective of this R21 proposal is to establish proof-of-concept for alterations in glucose homeostasis following intake of sucralose, but not aspartame, in middle-aged/older adults with prediabetes compared to a eucaloric diet with no NNS. We will investigate changes in inflammatory markers as potential mechanisms by which sucralose intake influences glucose homeostasis. Following a 2-week eucaloric lead-in diet, 30 middle-aged/older adults (40+ yrs) with prediabetes will be randomly assigned to 1 of 3 controlled feeding conditions for 6 weeks (10 participants per group): sucralose, aspartame, or a control group (no NNS). Standardized diets will be matched for macronutrients (50% carbohydrate, 35% fat, 15% protein) and other variables to avoid the potential confounds of weight change and dietary factors which may influence study outcomes (e.g., added sugars). All groups will receive identical diets, other than the additional NNS for the two NNS groups. 24-hr glycemic control using continuous glucose monitoring and insulin sensitivity and beta cell function via oral glucose tolerance test (OGTT), serum endotoxin, and inflammatory cytokines, including C-reactive protein, will be measured before and following the 6-week dietary treatment period. This research may have clinical practice and policy implications by informing U.S. dietary guidelines and guidelines for T2D prevention, which devote minimal attention to NNS and provide unclear guidance on NNS use due largely to a lack of rigorously-designed controlled feeding trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 40+ years
* Prediabetic (fasting glucose concentration of 100-125 mg/dL, 2-hour oral glucose tolerance test glucose concentration of 140-199 mg/dL, or a HbA1c value of 5.7% to 6.4%)
* Weight stable for previous 6 months (±2 kg)
* BMI <40 kg/m2
* Sedentary to recreationally active
* No plans to gain/lose weight or change physical activity level
* Willing to pick up food daily and consume foods provided for an 8-week period
* Verbal and written informed consent
* Approval by Medical Director
* Consume less than one serving of non-nutritive sweetener per week

Exclusion Criteria:

* BMI >40 kg/m2
* Diabetes or diabetes medication
* Antibiotic, prebiotic or prebiotic use in prior 3 months
* Uncontrolled hypertension (blood pressure (BP) > 159/99 mmHg)
* Diagnosed inflammatory bowel disease
* Past or current heart diseases, stroke, respiratory disease, endocrine or metabolic disease, or hematological-oncological disease
* Vegetarian or vegan
* Pregnant or plans to become pregnant
* Breastfeeding
* Food allergies or aversions, Phenylketonuria (PKU)
* Estrogen or testosterone usage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
24-hour glycemic control | 6 weeks
  The area under the curve (AUC) glucose concentrations, mg/dl from the continuous glucose monitoring at baseline and follow-up will be used

SECONDARY OUTCOMES:
Oral glucose tolerance | 6 weeks
  Oral glucose tolerance in response to 75 g glucose load; levels of glucose mg/dl will be determined 2 hrs after consuming a 75 glucose load
Insulin Sensitivity | 6 weeks
  Insulin uU/mL concentrations from the oral glucose tolerance test at baseline and follow-up will be used
Serum Endotoxin | 6 weeks
  Serum endotoxin mg/L concentrations will be measured at baseline and follow-up
C-reactive protein | 6 weeks
  C-reactive protein mg/dL concentrations will be measured at baseline and follow-up
Tumor Necrosis Factor alpha | 6 weeks
  Inflammatory cytokine: Tumor Necrosis Factor alpha pg/mL concentrations will be measured at baseline and follow-up
Interleukin 6 | 6 weeks
  Inflammatory cytokine: Interleukin 6 pg/mL concentrations will be measured at baseline and follow-up
Monocyte chemoattractant protein-1 | 6 weeks
  Inflammatory cytokine: Monocyte chemoattractant protein-1 pg/mL concentrations will be measured at baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Valisa Hedrick, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be posted to Virginia Tech's data repository, VTechData (https:// data.lib.vt.edu/). Datasets selected for sharing will be made accessible through VTechData, managed by the University Libraries at Virginia Tech. VTechData highlights, preserves, and provides access to data generated at Virginia Tech. The system relies on item/dataset level metadata as the primary building block to data discovery, access, and reuse. Published datasets are to be made accessible for at least five years.
Time Frame: Data will be available following completion of the trial and will be available for at least 5 years
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: http://data.lib.vt.edu/